CLINICAL TRIAL: NCT06820970
Title: Chronic Remote Ischemic Conditioning Combined With Mindfulness Therapy for Cardiovascular Adverse Events in Patients With Incomplete Revascularization of Coronary Artery Disease: A Multicenter, Double-blind, Randomized Controlled Trial
Brief Title: CRIC Combined With MFT for Cardiovascular Adverse Events in Patients With Incomplete Revascularization of CAD
Acronym: CRCMF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HenanICE202501
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This study adopts a 2×2 factorial randomized controlled trial design to evaluate the independent and combined effects of chronic remote ischemic preconditioning (CRIC) and mindfulness therapy (MFT) on anxiety and sleep quality in patients with coronary heart disease. Participants will be randomly assigned to one of four groups: (1) CRIC plus MFT, (2) CRIC only, (3) MFT only, or (4) neither intervention (control). The design allows the assessment of the main effects of RIPC and MBT, as well as the potential interaction effect between the two interventions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CRIC+MFT (Experimental): CIRC: Using a semi-automated machine, the pressure is increased according to the patient's own blood pressure level (20-40mmHg) when the cuff is pressed, and the pressure is compressed for 6 minutes per cycle, and the rest is 4 minutes per cycle.
  MFT: Participants receive guided mindfulness audio sessions twice daily for ~30 minutes each throughout the perioperative period. Content includes standardized mindfulness practices (e.g., focused attention, body awareness, nonjudgmental observation) designed to reduce anxiety and improve sleep quality.
  Interventions: Device: chronic remote ischemic conditioning; Behavioral: Mindfulness Therapy
- Control (neither CRIC nor MFT). (Sham Comparator): Sham CRIC: The pressure was 60mmHg when the cuff was pressurized, and the other modes were the same as in the CIRC group.
  Sham MFT: Health Education + Relaxation (HER): A time- and attention-matched audio program (twice daily, 30 minutes) delivering perioperative recovery and sleep-hygiene education with passive relaxation (music or simple muscle loosening), excluding mindfulness-specific techniques (no present-moment/nonjudgmental awareness training, no breath-focused meditation, no open monitoring).
  Interventions: Other: sham CRIC; Behavioral: sham MFT
- CRIC+sham MFT (Sham Comparator): CIRC: Using a semi-automated machine, the pressure is increased according to the patient's own blood pressure level (20-40mmHg) when the cuff is pressed, and the pressure is compressed for 6 minutes per cycle, and the rest is 4 minutes per cycle.
  Sham MFT-Health Education + Relaxation (HER): A time- and attention-matched audio program (twice daily, 30 minutes) delivering perioperative recovery and sleep-hygiene education with passive relaxation (music or simple muscle loosening), excluding mindfulness-specific techniques (no present-moment/nonjudgmental awareness training, no breath-focused meditation, no open monitoring).
  Interventions: Device: chronic remote ischemic conditioning; Behavioral: sham MFT
- Sham CRIC+MFT (Sham Comparator): Sham CRIC: The pressure was 60mmHg when the cuff was pressurized, and the other modes were the same as in the CIRC group.
  MFT: Participants receive guided mindfulness audio sessions twice daily for ~30 minutes each throughout the perioperative period. Content includes standardized mindfulness practices (e.g., focused attention, body awareness, nonjudgmental observation) designed to reduce anxiety and improve sleep quality.
  Interventions: Behavioral: Mindfulness Therapy; Other: sham CRIC

INTERVENTIONS:
Device: chronic remote ischemic conditioning — Using a semi-automated machine, the pressure is increased according to the patient's own blood pressure level (20-40mmHg) when the cuff is pressed, and the pressure is squeezed for 6 minutes per cycle and the rest is 4 minutes, for a total of 4 cycles per cycle.
  Other Names: CRIC
  Arms: CRIC+MFT; CRIC+sham MFT
Behavioral: Mindfulness Therapy — Participants receive guided mindfulness audio sessions twice daily for ~30 minutes each throughout the perioperative period. Content includes standardized mindfulness practices (e.g., focused attention, body awareness, nonjudgmental observation) designed to reduce anxiety and improve sleep quality.
  Other Names: MFT
  Arms: CRIC+MFT; Sham CRIC+MFT
Other: sham CRIC — The pressure was 60mmHg when the cuff was pressurized, and the other modes were the same as those of the CIRC group.
  Arms: Control (neither CRIC nor MFT).; Sham CRIC+MFT
Behavioral: sham MFT — Sham MFT: Health Education + Relaxation (HER): A time- and attention-matched audio program (twice daily, 30 minutes) delivering perioperative recovery and sleep-hygiene education with passive relaxation (music or simple muscle loosening), excluding mindfulness-specific techniques (no present-moment/nonjudgmental awareness training, no breath-focused meditation, no open monitoring).
  Arms: CRIC+sham MFT; Control (neither CRIC nor MFT).

SUMMARY:
The main objective of this study is to demonstrate whether the combination of chronic remote ischemic conditioning and mindfulness therapy can reduce cardiovascular adverse events in patients with incomplete revascularization of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old
* 2) Consistent with the diagnosis of coronary heart disease, complete revascularization was not performed (coronary angiography showed that at least one vessel with a reference diameter of 3.0mm had stenosis greater than 90%, and quantitative flow ratio (QFR) < 0.80)
* 3) Symptoms of myocardial ischemia (resting or exertional angina; Angina allele: chest tightness, shortness of breath, etc.);

Exclusion Criteria:

* Age < 18 years old
* Heart failure patients with NYHA class IV, or left ventricular ejection fraction (LVEF) < 30%
* Creatinine clearance <15 mL/min (or eGFR < 15 mL/min/1.73m²), or requires dialysis
* Myocardial diseases such as hypertrophic cardiomyopathy, dilated cardiomyopathy, etc.
* Uncontrolled or recurrent arrhythmic events (e.g., ventricular fibrillation, recurrent or symptomatic sustained ventricular tachycardia, complete heart block, atrial fibrillation with rapid ventricular rates, supraventricular tachycardia refractory to drugs)
* Poorly controlled hypertension (SBP > 180 mm Hg or DBP > 110 mm Hg)
* Active liver disease or persistent ALT or AST elevation ≥ 3 times the upper limit of normal
* Unexplained CK > 5 times the upper limit of normal, or elevated CK due to known muscle disease
* Planned or anticipated cardiac surgery or revascularization before randomization
* History of active malignancy (surgery, radiation therapy, and/or systemic therapy within the past 3 years)
* Diagnosed or suspected upper extremity vascular malformations, aneurysms, arteriovenous fistulas, or thrombosis
* Hearing impairment, unable to undergo mindfulness therapy
* Currently participating in another drug or device study, or within 30 days of completing another drug or device study or receiving another investigational drug
* Any life-threatening comorbid conditions expected to result in death within the next year (excluding cardiovascular diseases)
* Alcoholism, substance abuse history; and unwilling or unable to stop alcohol or substance abuse during the study
* History of major organ transplant (e.g., lung, liver, heart, bone marrow, kidney)
* Investigator's judgment of known major active and uncontrolled disease, or any medical, physical, or surgical conditions (e.g., infection, significant blood, kidney, metabolic, gastrointestinal, or endocrine dysfunction) that may interfere with participation in the clinical study
* As known to the investigator, the subject is unlikely to complete follow-up for more than 1 year or is expected to be unable to comply with the study requirements or understand the study's objectives and potential risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3420 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE | 12 months
  Clinical events were defined as: cardiac death, nonfatal myocardial infarction, hospitalization for new heart failure, hospitalization for angina pectoris

SECONDARY OUTCOMES:
Incidence of Cardiac Death | 3，6，9，12，24months
  Death is considered cardiac unless there is clear evidence of non-cardiac death
Incidence of Non-fatal Myocardial Infarction | 3，6，9，12，24months
  Includes STEMI and NSTEMI with elevated serum troponin on the basis of patient symptoms or ECG changes
Incidence of hospitalisation for new-onset heart failure | 3，6，9，12，24months
  New onset of heart failure-related symptoms with elevated serum BNP or NT-ProBNP
Incidence of hospitalised for angina pectoris | 3，6，9，12，24months
  Hospitalisation for angina pectoris symptoms of all causes, with a discharge diagnosis of angina pectoris
Incidence of unplanned revascularisation | 3，6，9，12，24months
  Unplanned revascularisation
Incidence of all cause death | 3，6，9，12，24months
  Death from any cause
Incidence of total length of hospitalization due to coronary heart disease | 3，6，9，12，24months
  Refers to the number of days when all hospitalizations for all causes of coronary heart disease are stacked together
Medical expenses due to coronary heart disease | 3，6，9，12，24months
  Refers to medical expenses incurred as a result of coronary heart disease
Degree of improvement in angina symptoms | 3，6，9，12，24months
  The degree of improvement in angina symptoms will be assessed using the Seattle Angina Questionnaire (SAQ), a 19-item self-administered questionnaire that evaluates five domains of health status in patients with coronary artery disease: physical limitation (9 items), angina stability (1 item), angina frequency (2 items), treatment satisfaction (4 items), and disease perception (3 items). Each domain score ranges from 0 to 100, with higher scores indicating better function (e.g., less physical limitation, less frequent angina, and better quality of life). A summary score, averaging the physical limitation, angina frequency, and quality of life domains, also ranges from 0 to 100. Improvement will be measured as the change in SAQ domain scores and summary score from baseline to follow-up time points, where an increase of 10 points or more in any domain or the summary score is considered clinically significant.
Change in anxiety scores | 3，6，9，12，24months
  Changes in anxiety scores will be assessed using the Zung Self-Rating Anxiety Scale (SAS), a 20-item self-report questionnaire that measures anxiety symptoms across cognitive, autonomic, motor, and central nervous system domains. Each item is rated on a 4-point Likert scale (1 = "none or a little of the time" to 4 = "most or all of the time"), yielding a raw total score ranging from 20 to 80, with higher scores indicating greater anxiety severity. Raw scores can be converted to an index score by multiplying by 1.25 (range: 25 to 100). The change in anxiety scores will be calculated as the difference in raw SAS scores from baseline to follow-up time points. For reference, raw scores are typically interpreted as: <36 (normal), 36-47 (mild anxiety), 48-59 (moderate anxiety), and ≥60 (severe anxiety).
Change in depression scores | 3，6，9，12，24months
  Changes in depression scores will be assessed using the Zung Self-Rating Depression Scale (SDS), a 20-item self-report questionnaire that measures depressive symptoms across affective, psychological, and somatic domains. Each item is rated on a 4-point Likert scale (1 = "none or a little of the time" to 4 = "most or all of the time"), yielding a raw total score ranging from 20 to 80, with higher scores indicating greater depression severity. Raw scores can be converted to an index score by multiplying by 1.25 (range: 25 to 100). The change in depression scores will be calculated as the difference in raw SDS scores from baseline to follow-up time points. For reference, raw scores are typically interpreted as: <40 (normal), 40-47 (mild depression), 48-55 (moderate depression), and ≥56 (severe depression).
Changes in sleep quality | 3，6，9，12，24months
  Changes in sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report questionnaire that evaluates sleep quality over the past month across seven components: subjective sleep quality (1 item), sleep latency (2 items), sleep duration (1 item), habitual sleep efficiency (3 items), sleep disturbances (9 items), use of sleeping medication (1 item), and daytime dysfunction (2 items). Each component is scored from 0 to 3, with higher scores indicating greater dysfunction. The global PSQI score is the sum of the seven components and ranges from 0 to 21, with higher scores indicating poorer sleep quality. Changes in sleep quality will be calculated as the difference in global PSQI scores from baseline to follow-up time points. For reference, a global score >5 is indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Muwei LI, MD, Study Chair — Fuwai Central China of Cardiovascular Hospital
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Main research content 2 years after the publication of the paper
Access Criteria: It is available on reasonable request from the contact person for the study